CLINICAL TRIAL: NCT01710176
Title: Localized High-Risk Soft Tissue Sarcomas Of The Extremities And Trunk Wall In Adults: An Integrating Approach Comprising Standard Vs Histotype-Tailored Neoadjuvant Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Italian Sarcoma Group (Network)
Collaborators: French Sarcoma Group (Other); Grupo Espanol de Investigacion en Sarcomas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISG-STS 10-01
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Localized High-risk Soft Tissue Sarcomas of the Extremities and Trunk Wall in Adults
MeSH Terms: interventions — Epirubicin; Ifosfamide; Gemcitabine; Docetaxel; Trabectedin; Etoposide; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard chemotherapy with full-dose epirubicin + ifosfamide (Active Comparator): Standard arm foresees 3 cycles of preoperative chemotherapy, each cycle will be repeated every 21 days and includes: epirubicin 60 mg/m2/day, short infusion, days 1 and 2; ifosfamide 3 g/m2/day, days 1, 2, 3
  Interventions: Drug: epirubicin 60 mg/m2/day (days 1, 2) and ifosfamide 3 g/m2/day (days 1, 2, 3)
- histotype-tailored chemotherapy according to the histotype (Experimental): gemcitabine+docetaxel for undifferentiated pleomorphic sarcoma, trabectedin for myxoid liposarcoma with hypercellularity, ifosfamide for synovial sarcoma, ifosfamide+etoposide for malignant peripheral nerve sheath tumor, gemcitabine+dacarbazine for leiomyosarcoma
  Interventions: Drug: gemcitabine 900 mg/m2 (days 1 and 8) and docetaxel 75 mg/m2 (day 8); Drug: trabectedin 1.3 mg/m2; Drug: high-dose ifosfamide 14 g/m2, given in in 14 days; Drug: etoposide 150 mg/m2/day (days 1, 2, 3) and ifosfamide 3g/m2/day (days 1, 2, 3); Drug: gemcitabine 1800 mg/m2 (day 1) and dacarbazine 500 mg/m2 (day 1)

INTERVENTIONS:
Drug: epirubicin 60 mg/m2/day (days 1, 2) and ifosfamide 3 g/m2/day (days 1, 2, 3)
  Arms: standard chemotherapy with full-dose epirubicin + ifosfamide
Drug: gemcitabine 900 mg/m2 (days 1 and 8) and docetaxel 75 mg/m2 (day 8)
  Arms: histotype-tailored chemotherapy according to the histotype
Drug: trabectedin 1.3 mg/m2
  Arms: histotype-tailored chemotherapy according to the histotype
Drug: high-dose ifosfamide 14 g/m2, given in in 14 days
  Arms: histotype-tailored chemotherapy according to the histotype
Drug: etoposide 150 mg/m2/day (days 1, 2, 3) and ifosfamide 3g/m2/day (days 1, 2, 3)
  Arms: histotype-tailored chemotherapy according to the histotype
Drug: gemcitabine 1800 mg/m2 (day 1) and dacarbazine 500 mg/m2 (day 1)
  Arms: histotype-tailored chemotherapy according to the histotype

SUMMARY:
This is a randomized Phase III clinical trial in the setting of localized high-risk soft tissue sarcomas (STS). This study will compare a standard neoadjuvant chemotherapy with epirubicin plus ifosfamide versus a histology-driven chemotherapy, i.e. a chemotherapy tailored to the specific histology within the family of adult STS. Chemotherapy will be administered for 3 cycles. There will be five histological groups (representing 80% of STS), as follows: leiomyosarcoma, myxoid liposarcoma with hypercellularity (round cell MLPS), synovial sarcoma, malignant peripheral nerve sheath tumor (MPNST) and undifferentiated pleomorphic sarcoma. The histology-driven chemotherapy for these groups will be, respectively, gemcitabine plus dacarbazine, trabectedin, high-dose ifosfamide, ifosfamide plus etoposide, gemcitabine plus docetaxel. Other histological groups will also be included and registered, but treated only by standard chemotherapy. Patients who have already undergone definitive surgery will receive treatment post-operatively and patients needing a re-excision after inadequate surgery will be treated as patients in the two groups, but of course will not be evaluable for response. A centralized pathological review will be performed. Radiological response will be evaluated according to RECIST and to Choi criteria. Pathological response will also be recorded.

The endpoint will be disease-free survival (DFS) and, secondarily, overall survival (OS) of patients receiving standard chemotherapy versus those receiving histotype-tailored chemotherapy. Additional aims will be to compare the probability of response of standard vs histotype-tailored chemotherapy and to determine the radiological and pathological response with standard chemotherapy vs tailored chemotherapy in each different histological group. Another aim will be to validate the response (both radiological and pathological) to preoperative chemotherapy as a surrogate endpoint for DFS and OS.

Three hundred patients will be randomized over a 3-years period, from a pool of 400-450 registered patients.

Translational research will be performed. Areas of research will include identification and validation of the potential predictive markers for each histological subgroups.

The study is designed to verify the statistical hypothesis that histotype-tailored approach is associated, overall, with a 30% reduction in the hazard of relapse. However, in each different histological group, the effect of histotype-tailored chemotherapy, as compared to standard chemotherapy, can be different. To address this weakness an orthogonal study of response to chemotherapy as a surrogate of DFS and OS has been introduced into the trial. This study intends to extensively investigate the response (radiological and pathological) to preoperative chemotherapy and to validate it as a surrogate endpoint by showing that it correlates with disease free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Soft tissue sarcoma of adults, primary or locally recurrent, with spindle-cell or pleomorphic histology, belonging to one of the following for the randomization (Group1):

   myxoid-Round Cell liposarcoma (cellular component >5 %), leiomyosarcoma, synovial sarcoma, malignant peripheral nerve sheat tumor, undifferentiated pleomorphic sarcoma (ex Malignant fibrous histiocytoma)

   Or belonging to one of the following for the registration (Group 2):

   myxofibrosarcoma, unclassified Spindle Cell, pleomorphic liposarcoma, pleomorphic rabdomiosarcoma Or belonging to either group but not being evaluable for response (re-excision after previous inadequate resection or primary definitive surgery) (Group3).

   The histological diagnosis must be made according to the WHO criteria and will have to be centrally reviewed before randomization.
2. High malignancy grade: grade 3 of 3, according to Coindre, or grade 2 at biopsy with a radiological evidence of more than 50% of necrosis in the tumor mass.
3. Deep seated extremities, girdles and/or superficial trunk (thoracic or abdominal wall)lesion.
4. Size of primary tumor (visible or previously inadequately resected) >5 cm at instrumental staging (CT, MRI), or locally recurrent of any size.
5. Age > 18 years.
6. ECOG performance status <1.
7. Adequate bone marrow function:

   WBC >3.500/mm3 neutrophil >1.500/mm3 platelets >150.000/mm3 hemoglobin >11 g%.
8. Adequate renal (creatinine <1.3 mg%), and hepatic function (bilirubin <1.5 mg% and transaminases <2 x n.v. If ALP > 2.5 x ULN, ALP LF and/or GGT < ULN).
9. Adequate cardiac function (FE >50%).
10. Signed informed consent.
11. Complete compliance of the participating center with the protocol requirements.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Distant metastasis.
3. Other malignancies within past 5 years, with the exception of carcinoma in situ of cervix and basocellular skin cancers treated with eradicating intent.
4. Sarcoma histotypes other than those mentioned in the inclusion criteria.
5. Prior CT and/or RT.
6. Serious psychiatric disease that precludes informed consent or limits compliance.
7. Medical disease limiting survival to less than two years, limiting compliance or which in the physician's opinion might interfere significantly with the toxicity of the treatments.
8. Cardiovascular diseases resulting in a New York Heart Association Functional Status > 2.
9. Uncontrolled bacterial, viral or fungal infection.
10. Impossibility of ensuring adequate follow-up.
11. Failure to comply with the requirements of the present protocol leading to exclusion of the participating center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
To compare the effect on disease-free survival of full-dose standard chemotherapy with histotype-tailored chemotherapy within the context of an integrated strategy for high risk soft tissue sarcomas typical of the adult. | 5 years

SECONDARY OUTCOMES:
1:overall survival 2:response in the whole population 3:response by RECIST and Choi in each different histotype 4:pathological response 5:feasibility of integration of preoperative chemotherapy with preoperative local-regional treatments 6:PET re | 5 years

OTHER OUTCOMES:
To validate the response to preoperative chemotherapy (both radiological and pathological) as a surrogate endpoint by showing that disease free survival and overall survival depend on response status and are independent of the treatment arm. | 5 years

CONTACTS AND LOCATIONS:
Locations (15):
- Italy (12):
  - Fondazione Del Piemonte Per L'Oncologia Ircc Di Candiolo -, Candiolo, TO
  - Irccs Centro Di Riferimento Oncologico (Cro) -, Aviano (PN)
  - Irccs Istituto Ortopedico Rizzoli (Ior) -, Bologna
  - Pres.Ospedal.Spedali Civili Brescia -, Brescia
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori -, Meldola (FC)
  - Irccs Istituto Europeo Di Oncologia (Ieo) -, Milan
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan
  - Irccs Istituto Nazionale Tumori Fondazione Pascale -, Napoli
  - Irccs Istituto Oncologico Veneto (Iov), Padua
  - Irccs Istituto Regina Elena (Ifo), Roma
  - Irccs Istituto Clinico Humanitas -, Rozzano (MI)
  - Presidio Sanitario Gradenigo Di Torino, Torino
- Spain (3):
  - Hospital Vall D'Hebron, Barcelona
  - Hospital Clínico de Malaga, Málaga
  - Hospital Son Espases, Palma de Mallorca

REFERENCES:
- [Derived] Gronchi A, Palmerini E, Quagliuolo V, Martin Broto J, Lopez Pousa A, Grignani G, Brunello A, Blay JY, Tendero O, Diaz Beveridge R, Ferraresi V, Lugowska I, Pizzamiglio S, Verderio P, Fontana V, Donati DM, Palassini E, Sanfilippo R, Bianchi G, Bertuzzi A, Morosi C, Pasquali S, Stacchiotti S, Bague S, Coindre JM, Miceli R, Dei Tos AP, Casali PG. Neoadjuvant Chemotherapy in High-Grade Myxoid Liposarcoma: Results of the Expanded Cohort of a Randomized Trial From Italian (ISG), Spanish (GEIS), French (FSG), and Polish Sarcoma Groups (PSG). J Clin Oncol. 2024 Mar 10;42(8):898-906. doi: 10.1200/JCO.23.00908. Epub 2024 Jan 17. PMID 38232337
- [Derived] Gronchi A, Palmerini E, Quagliuolo V, Martin Broto J, Lopez Pousa A, Grignani G, Brunello A, Blay JY, Tendero O, Diaz Beveridge R, Ferraresi V, Lugowska I, Merlo DF, Fontana V, Marchesi E, Braglia L, Donati DM, Palassini E, Bianchi G, Marrari A, Morosi C, Stacchiotti S, Bague S, Coindre JM, Dei Tos AP, Picci P, Bruzzi P, Casali PG. Neoadjuvant Chemotherapy in High-Risk Soft Tissue Sarcomas: Final Results of a Randomized Trial From Italian (ISG), Spanish (GEIS), French (FSG), and Polish (PSG) Sarcoma Groups. J Clin Oncol. 2020 Jul 1;38(19):2178-2186. doi: 10.1200/JCO.19.03289. Epub 2020 May 18. PMID 32421444
- [Derived] Gronchi A, Ferrari S, Quagliuolo V, Broto JM, Pousa AL, Grignani G, Basso U, Blay JY, Tendero O, Beveridge RD, Ferraresi V, Lugowska I, Merlo DF, Fontana V, Marchesi E, Donati DM, Palassini E, Palmerini E, De Sanctis R, Morosi C, Stacchiotti S, Bague S, Coindre JM, Dei Tos AP, Picci P, Bruzzi P, Casali PG. Histotype-tailored neoadjuvant chemotherapy versus standard chemotherapy in patients with high-risk soft-tissue sarcomas (ISG-STS 1001): an international, open-label, randomised, controlled, phase 3, multicentre trial. Lancet Oncol. 2017 Jun;18(6):812-822. doi: 10.1016/S1470-2045(17)30334-0. Epub 2017 May 9. PMID 28499583
- [Derived] Gronchi A, Stacchiotti S, Verderio P, Ferrari S, Martin Broto J, Lopez-Pousa A, Llombart-Bosch A, Dei Tos AP, Collini P, Jurado JC, De Paoli A, Donati DM, Poveda A, Quagliuolo V, Comandone A, Grignani G, Morosi C, Messina A, De Sanctis R, Bottelli S, Palassini E, Casali PG, Picci P. Short, full-dose adjuvant chemotherapy (CT) in high-risk adult soft tissue sarcomas (STS): long-term follow-up of a randomized clinical trial from the Italian Sarcoma Group and the Spanish Sarcoma Group. Ann Oncol. 2016 Dec;27(12):2283-2288. doi: 10.1093/annonc/mdw430. Epub 2016 Oct 11. PMID 27733375
- [Derived] Palassini E, Ferrari S, Verderio P, De Paoli A, Martin Broto J, Quagliuolo V, Comandone A, Sangalli C, Palmerini E, Lopez-Pousa A, De Sanctis R, Bottelli S, Libertini M, Picci P, Casali PG, Gronchi A. Feasibility of Preoperative Chemotherapy With or Without Radiation Therapy in Localized Soft Tissue Sarcomas of Limbs and Superficial Trunk in the Italian Sarcoma Group/Grupo Espanol de Investigacion en Sarcomas Randomized Clinical Trial: Three Versus Five Cycles of Full-Dose Epirubicin Plus Ifosfamide. J Clin Oncol. 2015 Nov 1;33(31):3628-34. doi: 10.1200/JCO.2015.62.9394. Epub 2015 Sep 8. PMID 26351345